CLINICAL TRIAL: NCT04127981
Title: A Pilot Bioimaging Trial of Cancer Cachexia
Brief Title: Medical Imaging of Cachexia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Olivia Newton-John Cancer Research Institute (Other)
Collaborators: La Trobe University (Other); Austin Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ONJ2018-002
Record Dates: First submitted 2019-04-23; First posted 2019-10-16 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Cancer Cachexia
Keywords: 18F-FDG PET Scan; Dexa Scan; Quality of Life assessment tools
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Intervention Model Description: 20 patients with advanced/metastatic colorectal, non-small cell lung cancer (NSCLC) or pancreatic cancer without cachexia, and 20 patients with advanced/metastatic colorectal, non-small cell lung cancer (NSCLC), or pancreatic cancer with documented cachexia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with cancer cachexia (Active Comparator): 20 patients with advanced/metastatic colorectal, non-small cell lung cancer (NSCLC), or pancreatic cancer with documented cachexia.
  Interventions: Diagnostic Test: 18F-FDG PET + Dexa Scan
- Patients without cancer cachexia (Active Comparator): 20 patients with advanced/metastatic colorectal, non-small cell lung cancer (NSCLC) or pancreatic cancer without cachexia.
  Interventions: Diagnostic Test: 18F-FDG PET + Dexa Scan

INTERVENTIONS:
Diagnostic Test: 18F-FDG PET + Dexa Scan — 18F-FDG PET will be compared with Dexa Scan result within and between arms.

SUMMARY:
This is a pilot trial using 18F-FDG PET and DXA scans to determine whether these investigations are objective tools to assess cachexia.

DETAILED DESCRIPTION:
This pilot study will establish the differences in BAT uptake of 18F-FDG in cachectic and non-cachectic cancer patients using PET imaging.

Patients willbe assessed for sarcopenia using a dual energy X-ray absorptiometry or bone densitometry scan (DXA). Given the variables which may affect uptake of BAT in cancer patients, this study will standardise patient preparation and PET scan procedure in order to obtain the most reliable assessment of BAT activity in all patients on study.

It is hypothesisd that use of this PET imaging technique, which is part of standard care to assess cancer progression, may assist clinicians in early identification of metabolic changes in a patient, with potential for early intervention and utility in monitoring success of treatments of cachexia.

A total of 40 patients will be evaluated, 20 patients with advanced/metastatic colorectal, non-small cell lung cancer (NSCLC) or pancreatic cancer without cachexia, and 20 patients with advanced/metastatic colorectal, non-small cell lung cancer (NSCLC), or pancreatic cancer with documented cachexia, all of whom are referred for standard of care 18F-FDG PET scans.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant disease;
* ECOG Performance score of 0-2;
* Age ≥ 18 years;
* Life expectancy of >4 months at screening;
* Cachexia patient group only: Fulfils diagnostic criteria for cachexia: unintentional weight loss more than 5% over the previous 6 months, or more than 2% in individuals with a decreased body-mass index of <20kg/m2, or skeletal muscle wasting (sarcopenia).

Exclusion Criteria:

Patients with uncontrolled Diabetes Mellitus;

* Psychological unstable persons presumed unfit to perform the investigations;
* Persons unable to lie or sit still for 1-2 hours;
* Pregnant patients;
* Patients who received high doses of radiotherapeutic radiation of the neck and/or upper chest in their medical history limiting nutritional intake;
* Patients who are receiving any chemotherapeutic agents which is limiting nutritional intake;
* Persons that received cervical or thoracic sympathectomy or have a nerve dysfunction which is likely to influence sympathetic nerves;
* The use of medication that influences the sympathetic nerve system: ß-blockers, α-blockers, central anti-hypertensives, certain anti-depression drugs (MAO inhibitors, tricyclic antidepressives), reserpine, cocaine, calcium channel blockers, labetalol, and certain tranquillizers (fenothiazines).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2023-12-28 (Estimated); Study Completion 2023-12-28 (Estimated)

PRIMARY OUTCOMES:
Correlation of a clinical diagnosis of cachexia with the metabolic activity of brown adipose tissue, bone density and muscle mass. | 7 days post enrollment
  Quantitation of the metabolic activity of brown adipose tissue, bone density and muscle mass using 18F-FDG uptake and bone densitometry will be correlated with a diagnosis of clinical cachexia.

SECONDARY OUTCOMES:
Optimization of PET scanning methods for imaging of brown adipose tissue. | 7 days post enrollment
  Optimization of the patient environment (ie. ambient temperature) and metabolic state (ie. Heart rate, dietary state) to minimize the impact of these factors and allow direct comparison of metabolic activity of brown adipose tissue between cachectic and non-cachectic patients.
To quantify change from normal of inflammatory blood biomarkers | 7 days post enrollment
  To validate change from normal laboratory range of inflammatory blood based proteins and enzymes in cachectic vs non-cachectic patients.
To quantify change from normal of immune blood biomarkers | 7 days post enrollment
  To validate change from normal laboratory range immune blood based proteins and enzymes in cachectic vs non-cachectic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Scott, MD, Principal Investigator — Austin Health/ONJCRI
Locations (1):
- Austin Health, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Cohort data will be shared via journal and conference presentations